CLINICAL TRIAL: NCT04570644
Title: A Phase I/II Randomized, Open-Labeled Study to Evaluate Pharmacokinetic and Pharmacodynamic Effects and Safety of ALZT-OP1 in Subjects With Alzheimer's Disease and Normal Healthy Volunteers
Brief Title: Randomized I/II Phase Study of ALZT-OP1 Combination Therapy in Alzheimer's Disease and Normal Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AZTherapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AZT-008
Record Dates: First submitted 2020-09-17; First posted 2020-09-30 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2020-09

CONDITIONS: Healthy Volunteers; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Cromolyn Sodium; Ibuprofen

STUDY DESIGN:
Intervention Model Description: ALZT-OP1a (cromolyn) and ALZT-OP1b (Ibuprofen) are being evaluated in this study.
Masking Description: A Phase I/ II Randomized, Open-Label Study to Evaluate Pharmacokinetic and Pharmacodynamic Effects and Safety of ALZT-OP1 (co-administration of ALZT-OP1a and ALZT-OP1b) in Subjects with Alzheimer's Disease and Normal Healthy Volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A (Other): 24 subjects randomized to receive treatment: (A-B) = Single 17.1 mg oral inhaled dose of ALZT-OP1a (cromolyn) via dry powder inhaler and a single oral 10 mg tablet of ALZT-OP1b (ibuprofen) on Day 1. On Day 2, subjects would receive two 17.1 mg doses of ALZT-OP1a via dry powder inhaler and two 10 mg tablets of ALZT-OP1b (ibuprofen), within two minutes of each other.
  (B-A) = Two 17.1 mg doses of ALZT-OP1a (cromolyn) and two doses of 10 mg ALZT-OP1b (ibuprofen) on Day 1 and single 17.1 mg dose of ALZT-OP1a cromolyn 17.1 mg and a single 10 mg dose of ALZT-OP1b (ibuprofen) on Day 2.
  All subjects will have plasma and CSF collected for PK analysis.
  Interventions: Drug: ALZT-OP1 (cromolyn and ibuprofen) ALZT-OP1a (cromolyn) and ALZT-OP1b (ibuprofen)
- Part B (Other): PD - 32 subjects (AD only) will be enrolled in the PD portion of the study. Twenty-four (24) subjects will be assigned to Treatment Group 1 to receive a single (17.1 mg) inhaled dose of ALZT-OP1a (cromolyn) plus a single (10 mg) oral dose of ALZT-OP1b (ibuprofen) daily for 60 days.
  All subjects will have plasma and CSF collected for PD biomarker analysis. Eight (8) A subjects will be assigned to Treatment Group 2 (Control Group) and will not be administered study drug.
  Interventions: Drug: ALZT-OP1 (cromolyn and ibuprofen) ALZT-OP1a (cromolyn) and ALZT-OP1b (ibuprofen)

INTERVENTIONS:
Drug: ALZT-OP1 (cromolyn and ibuprofen) ALZT-OP1a (cromolyn) and ALZT-OP1b (ibuprofen) — Drug : ALZT-OP1a
  1. Mast cell stabilizer
  2. Neuroinflammatory microglial modulator
  ALZT-OP1b anti-inflammatory
  Device: Dry Powder Inhaler The inhaler will be used to deliver ALZT-OP1a via oral inhalation for dosing on study.
  Other Names: Cromolyn, Intal, Cromolyn Sodium, Sodium cromoglycate; Ibuprofen

SUMMARY:
This is a randomized, open-label, cross-over, pharmacokinetic and pharmacodynamic PK/PD study. (Part A)The PK portion of the study is designed to evaluate the pharmacokinetics of ALZT-OP1 (a combination drug therapy) designated as ALZT-OP1a and ALZT-OP1b, in both plasma and CSF, following co-administration of the two active investigational products, in healthy volunteers and Alzheimer subjects aged 55-79 and in good health. (Part B) The PD portion of the study will evaluate the pharmacodynamics of ALZT- OP1, using both plasma and CSF biomarkers, following 60 days of consecutive daily treatment, in AD subjects only.

DETAILED DESCRIPTION:
This is a phase I/II randomized, open-label, cross-over, PK/PD study. The PK (Part A) portion of the study is designed to evaluate both single and double doses of ALZT-OP-1a (17.1mg or 34.2 mg) and ALZT-OP1b (10 mg or 20 mg) in both Alzheimer's subjects and healthy volunteers. The PD (Part B) portion of the study is designed to evaluate single doses of ALZT-OP-1a (17.1mg) and ALZT-OP1b (10 mg) in AD subjects treated for 60 days. An Alzheimer's control group will be utilized for comparison to active treatment groups but will not be administered study treatment; however, they will have biomarkers collected.

PK (Part A) n=24, both healthy volunteers and AD subjects

Part A is an open-label study, cross-over, PK study where 24 subjects will be randomly assigned to receive treatment regimen A-B or B-A for two consecutive day of dosing.

Subjects will be admitted to the Phase 1 unit the morning before dosing and will initiate dosing the following morning for 2 consecutive days of dosing (A-B, or B-A).

Day 1 (A-B) will consist of a single inhaled oral dose of ALZT-OP1a via dry powder inhaler + a single oral tablet dose of ALZT-OP1b.

Day 2 (B-A) will consist of two oral inhaled doses of ALZT-OP1a, not more than 2 mins apart, via dry powder inhaler + two oral tablets doses of ALZT-OP1b.

Day 1 (B-A) will consist of two oral inhaled doses of ALZT-OP1a, not more than 2 mins apart, via dry powder inhaler + two oral tablets doses of ALZT-OP1b.

Day 2 (A-B) regimen consists of a single inhaled oral dose of ALZT-OP1a via dry powder inhaler + a single oral tablet dose of ALZT-OP1b.

AD subjects will be given the option to roll over into the PD portion of the study.

PD (Part B) n=32, AD subjects only

Part B is an open-label, PD study where 32 AD subjects will be randomly assigned to receive either active treatment or be assigned to a non-treatment control arm.

Twenty-four (24) subjects will be randomly assigned to Treatment Group 1 to receive a single (17.1 mg) inhaled dose of ALZT-OP1a plus a single (10 mg) oral dose of ALZT-OP1b daily for 60 days.

Eight (8) subjects will be randomly assigned to Treatment Group 2 (Control Group) and will not be administered study drug.

All subjects will have plasma collected on Day 1, Day 30, and Day 60 and CSF collected on Day 1 and Day 60.

ELIGIBILITY:
Inclusion Criteria:

* For All Subjects

  1. Provide a signed written informed consent;
  2. Age 55-79 old (inclusive);
  3. ECG without abnormal, clinically significant findings;
  4. Body mass index (BMI) ≥ 18 kg/m2 and ≤ 30 kg/m2
  5. Negative urine drug screen for selected drugs of abuse at screening;
  6. Negative for hepatitis and HIV at screening;
  7. Negative for COVID-19 at screening;
  8. Good general health, as determined by medical history, physical examination, and clinical laboratory testing;
  9. Must provide written informed consent for CSF sampling. For AD Subjects Only

     In addition to satisfying all of the above inclusion criteria, AD subjects must also meet the following criteria:
  10. Diagnosed with mild to moderate Alzheimer's disease;
  11. Clinical Dementia Rating (Global) 0.5
  12. Mini-mental state examination (MMSE) ≤ 22;
  13. Must be fluent in the language of the cognitive testing material being administered;
  14. Stability of permitted medications for 4 weeks prior to study start;
  15. Visual and auditory acuity adequate for neuropsychological testing.
  16. Must provide written informed consent for APOe4 genotype testing; For All Subjects in Part A (PK)
  17. Willingness to stay in the unit overnight for the duration of the PK portion of the study.

Exclusion Criteria:

* For All Subjects

  1. Current smokers, or ex-smokers with a remote history (> 100 pack/year);
  2. Clinically significant medical conditions;
  3. History of abnormal clinically significant ECG abnormalities;
  4. Symptomatic viral infection, or suspicion thereof (including rhinitis) in the last 14 days prior to dosing;
  5. Signs of active pulmonary infection or other pulmonary inflammatory conditions, even in absence of febrile episodes, in the last 14 days;
  6. History or presence of disease in the kidneys and/or heart, lungs, liver, gastrointestinal tract, endocrine organs or other conditions such as metabolic disease known to interfere with the absorption, distribution, metabolism, and excretion of drugs;
  7. Malignancy, regardless of location;
  8. Autoimmune disorders such as (but not limited to) lupus erythematosus, multiple sclerosis, rheumatoid arthritis, or sarcoidosis;
  9. Investigational agents are prohibited one month prior to entry and for the duration of the trial;
  10. Currently taking medications known to be CYP2C9 inducers (e.g., carbamazepine and rifampicin;
  11. Currently taking cromolyn, or have taken cromolyn products, within the past 30 days;
  12. Non-steroidal anti-inflammatory drug (NSAID) use (products containing ibuprofen while on study);
  13. Allergy or hypersensitivity to cromolyn (also known as Intal®, Nasalcrom®, Opticrom®, Gastrocrom®, etc.);
  14. Allergy or hypersensitivity to ibuprofen (Advil®, Motrin®, Nuprin®, etc.) or aspirin, including Stevens-Johnson syndrome;
  15. History of hypersensitivity or allergies to any of the drug compound under investigation (cromolyn sodium, ibuprofen, lactose, or magnesium stearate);
  16. Current respiratory disorders and chronic respiratory disease with impaired respiratory effort or difficulty taking inhaled drugs (examples: COPD, emphysema);
  17. Abnormal pulmonary function test, defined for this protocol as: FEV1 < 70% of predicted value, indicating moderate or severe respiratory impairment;
  18. Any other disease or condition, which, in the opinion of the investigator, would make the subject unsuitable for this study;
  19. Female subjects of reproductive potential with a positive pregnancy test (urine or serum) or who are pregnant or lactating.

      For AD Subjects Only

      In addition to not meeting any of the above exclusion criteria for Normal Healthy Volunteers, AD subjects must also not meet any of the following criteria:
  20. Any significant neurological disease other than suspected incipient AD, such as Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities;
  21. Major depressive episode, as described in the Diagnostic and Statistical Manual of Mental Disorders (DSM-V) within the past 6 months, which could lead to difficulty complying with the protocol;
  22. History of schizophrenia or bipolar disorder (DSM-V criteria);
  23. Currently taking medications that could lead to difficulty complying with the protocol; For All Subjects in Part A (PK)
  24. Aspirin, or products containing aspirin, while on PK study; For All Subjects in Part B (PD)
  25. Chronic daily use of aspirin exceeding standard of care guidelines for low dose aspirin therapy for prevention of stroke and/or other recommended uses, while on PD study.

Ages: 55 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-01-18 (Actual)

PRIMARY OUTCOMES:
Part A Non-compartmental PK parameters will be calculated and reported for ALZT-OP1a and ALZT-OP1b | • 2 Days
  • PK profile for ALZT-OP1a and ALZT-OP1b in plasma and CSF
PK profile for ALZT-OP1a and ALZT-OP1b in plasma and CSF AUC 0-∞ | 2 Days
  Evaluation AUC 0-∞ (area under the curve from 0 to infinity)
PK profile for ALZT-OP1a and ALZT-OP1b in plasma and CSF AUC 0-t | 2 Days
  Evaluation AUC 0-t (area under the curve from 0 to t hours where t is the last measured concentration)
PK profile for ALZT-OP1a and ALZT-OP1b in plasma and CSF AUCPLASMA/AUCCSF | 2 Days
  Evaluation AUCPLASMA/AUCCSF (ratio at 60 min, 120 min, 240 min, 360 min and 480 min)
PK profile for ALZT-OP1a and ALZT-OP1b in plasma and CSF CL/F | 2 Days
  Evaluation CL/F (apparent total body clearance)
PK profile for ALZT-OP1a and ALZT-OP1b in plasma and CSF Cmax | 2 Days
  Evaluation Cmax (maximum plasma and CSF concentration observed)
PK profile for ALZT-OP1a and ALZT-OP1b in plasma and CSF t½ (half-life) | 2 Days
  Evaluation t½ (half-life)
PK profile for ALZT-OP1a and ALZT-OP1b in plasma and CSF tmax | 2 Days
  Evaluation tmax (sampling time at which Cmax occurred)
PK profile for ALZT-OP1a and ALZT-OP1b in plasma and CSF Vd/F | 2 Days
  Evaluation Vd/F (apparent volume of distribution)

SECONDARY OUTCOMES:
Biomarker Beta Amyloid (Αβ-42) Sample Analysis plasma and CSF Day 1 to 60 Days | Day 1 to Day 60
  Evaluation Beta Amyloid (Αβ-42)
Biomarker Beta Amyloid (Αβ-40) Sample Analysis plasma and CSF Day 1 to 60 Days | Day 1 to Day 60
  Evaluation Beta Amyloid (Αβ-40)
Biomarker Beta Amyloid (Αβ-38) Sample Analysis plasma and CSF Day 1 to 60 Days | Day 1 to Day 60
  Evaluation Beta Amyloid (Αβ-38)
Biomarker Total Tau Sample Analysis plasma and CSF Day 1 to 60 Days | Day 1 to Day 60
  Evaluation Total Tau
Biomarker Neurofilament light (Nf-L) Sample Analysis plasma and CSF Day 1 to 60 Days | Day 1 to Day 60
  Evaluation Neurofilament light (Nf-L)
Biomarker Glial Fibrillary Acidic Protein (GFAP) Sample Analysis plasma and CSF Day 1 to 60 Days | Day 1 to Day 60
  Evaluation Glial Fibrillary Acidic Protein (GFAP)
Biomarker P-Tau (Thr 231) Sample Analysis plasma and CSF Day 1 to 60 Days | Day 1 to Day 60
  Evaluation P-Tau (Thr 231)
Biomarker Interferon-γ (IFN-γ) Sample Analysis plasma and CSF Day 1 to 60 Days | Day 1 to Day 60
  Evaluation Interferon-γ (IFN-γ)
Biomarker Tumor Necrosis Factor-α (TNF-α) Sample Analysis plasma and CSF Day 1 to 60 Days | Day 1 to Day 60
  Evaluation Tumor Necrosis Factor-α (TNF-α)
Biomarker Transforming Growth Factor-β1 (TGF-β1) Sample Analysis plasma and CSF Day 1 to 60 Days | Day 1 to Day 60
  Evaluation Transforming Growth Factor-β1 (TGF-β1)
Biomarker CD33 Sample Analysis plasma and CSF Day 1 to 60 Days | Day 1 to Day 60
  Evaluation CD33
Biomarker Triggering Receptor Expressed on Myeloid Cells-2 (TREM2) Sample Analysis plasma and CSF Day 1 to 60 Days | Day 1 to Day 60
  Evaluation Triggering Receptor Expressed on Myeloid Cells-2 (TREM2)
Biomarker Neurogranin Sample Analysis plasma and CSF Day 1 to 60 Days | Day 1 to Day 60
  Evaluation Neurogranin

OTHER OUTCOMES:
Number of Treatment Emergent Adverse Events (TEAE) | 2 Days Part A and 60Days Part B
  Safety will be evaluated based on the number, type, and frequency of treatment emergent adverse events. They will be individually presented for all subjects in data listings, and summarized in tables by treatment group and by treatment assignment. The AEs will be summarized and reported collectively based on information obtained through physical examination, ECG, and laboratory findings captured after dosing was initiated.

CONTACTS AND LOCATIONS:
Overall Officials: David R. Elmaleh, PhD, Study Chair — AZTherapies, Inc.
Locations (1):
- Panax Clinical Research, Miami Lakes, Florida, United States

REFERENCES:
- See also: Pharmacokinetics of Cromolyn and Ibuprofen in Healthy Elderly Volunteers — https://link.springer.com/article/10.1007/s40261-017-0549-5